CLINICAL TRIAL: NCT03354741
Title: Stimulation of Acupuncture Points by Athermic Laser Therapy for the Prevention of Chemotherapy Induced Nausea and Vomiting in Children
Acronym: NAUVOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17-AOI-06
Record Dates: First submitted 2017-11-08; First posted 2017-11-28 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-09

CONDITIONS: Children; Chemotherapy-induced Nausea and Vomiting; Malignant Tumor
MeSH Terms: conditions — Vomiting; Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser then Sham therapy (Other): 2nd cycle of chemotherapy : administration of laser therapy 3th cycle of chemotherapy : administration of a sham laser according to the same modalities
  Interventions: Other: laser therapy
- Sham therapy then laser (Other): 2nd cycle of chemotherapy : administration of a sham laser 3th cycle of chemotherapy : administration of laser therapy according to the same modalities
  Interventions: Other: laser therapy

INTERVENTIONS:
Other: laser therapy — stimulation of the acupuncture point P6 by laser therapy

SUMMARY:
Poor control of chemotherapy-induced nausea and vomiting has a major clinical and psychological impact in patients treated with chemotherapy. Metabolic, nutritional and mechanical complications, as well as psychological repercussions, complicate the therapeutic management of the patient and can lead to poor compliance, a deterioration in the general condition or even prolongation of hospitalizations and a delay in the implementation of chemotherapy cures. The control of induced chemo- and radio-induced nausea and vomiting rests above all on their prevention. At present and in most centers, the prevention of nausea and vomiting in the pediatric onco-hematology department of the CHU de Nice is based exclusively on drug treatments, according to a protocol established according to the emetogenic risk of the chemotherapy received.

We propose a study evaluating the effectiveness of the stimulation of acupuncture points by low frequency laser therapy associated with antiemetics in the management of chemotherapy induced nausea and vomiting in patients of 2 to 20 years followed in the service of analgesics. pediatric onco-hematology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant pathology with indication of chemotherapy with moderate to severe emetogenic potential
* Indication of at least three identical chemotherapy cures
* Age between 2 and 20 years
* Prescription of an anti emetic protocol
* Karnosky / Lansky Index> 60%

Exclusion Criteria:

* Proven laser contraindication
* Vomiting in the 24 hours before starting treatment
* Presenting a brain lesion responsible for nausea and vomiting
* Pelvic abdominal irradiation the week before the start of treatment
* Treatment with benzodiazepines or opioids the week before treatment
* Pregnant women

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
The complete response to the preventive treatment of nausea and vomiting | Hours 72 after the end of chemotherapy
  The complete response to the preventive treatment of nausea and vomiting defined by the absence of vomiting (active rejection by the mouth of part of the contents of the stomach), absence of nausea (effort of vomiting without active rejection) and the lack of emergency antiemetic treatment during the acute and delayed phase of chemotherapy (from the onset of chemotherapy to H72 after the end of chemotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyne POIREE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Dr Marilyne POIREE, Nice, France

IPD SHARING:
Plan to Share IPD: No